CLINICAL TRIAL: NCT00924092
Title: Open Label Phase I Study to Evaluate the Safety and Tolerability of Vaccine (GI-6207) Consisting of Whole, Heat-Killed Recombinant Saccharomyces Cerevisiae Genetically Modified to Express CEA Protein in Adults With Metastatic CEA-Expressing Carcinoma
Brief Title: An Open Label Phase I Study to Eval the Safety and Tolerability of a Vaccine (GI-6207) Consisting of Whole, Heat-killed Recombinant Saccharomyces Cerevisiae (Yeast) Genetically Modified to Express CEA Protein in Adults With Metastatic CEA-expressing ...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090101; 09-C-0101; NCT00887016 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2014-05-20

CONDITIONS: Prostate Cancer; Breast Cancer; Lung Cancer; Colorectal Cancer; Head and Neck Cancer
Keywords: Immunotherapy; Lung Cancer; Colorectal Cancer; Head and Neck Cancer; Prostate; Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms | interventions — yeast-CEA vaccine

INTERVENTIONS:
Biological: GI-6207 [Recombinant Saccharomyces Cerevisia
Drug: (Yeast CEA Vaccine)(GI-6207[Recombinant Sarrcharomyces Cerevusua-CEA (610D)])

SUMMARY:
Objectives:

* To find out the maximum tolerated dose of the GI-6207 vaccine (the highest dose that does not cause unacceptable side effects), and to evaluate any side effects.
* To see if GI-6207 has any effect on patients tumors.
* To learn how the vaccine causes immune responses against the cancer.

Eligibility:

* Patients 18 years of age and older who have been diagnosed with a cancer that has not responded to standard treatments. Patients must not be allergic to yeast or yeast products.

Design:

* Initial physical examination, blood and tissue sampling, computed tomography (CT) scan, and skin test to determine eligibility for the procedure.
* Treatment with GI-6027 in seven 14-day cycles as follows:
* Vaccine administered on days 1, 15, 29, 43, 57, 71, and 85.
* Vaccine given at four sites around the body: right and left chest area below the armpit, and right and left upper thigh in the pelvic region. (These areas drain into parts of your body that contain large numbers of lymph nodes. The lymph nodes contain immune cells that may be activated by the vaccine to target cancer cells.)
* Clinic visits for physical examinations to check vital signs, take additional blood and urine samples, and perform other tests needed for the study.
* After day 85 (about 3 months), patients will continue to receive vaccine monthly (or every 28 days) as long as the vaccine is not producing harmful effects or side effects and the cancer is either stable or reducing. Patients who do well on the vaccine may continue to receive it for as long as it is available.

DETAILED DESCRIPTION:
Background:

Carcinoembryonic antigen (CEA) is overexpressed in multiple adenocarcinomas.

Previous clinical studies utilizing CEA-based vaccine therapy have demonstrated safety, T-cell immune responses against CEA, and preliminary evidence of clinical benefit.

Preclinical studies have shown that Saccharomyces-CEA (yeast-CEA) can induce a strong immune response to CEA as well as therapeutic antitumor responses in a CEA-transgenic host.

Previous and ongoing clinical studies utilizing whole, heat-killed recombinant Saccharomyces cerevisiae yeast genetically modified to express mutated Ras (GI-4000) or hepatitis C (GI-5005) proteins demonstrated this vaccine vehicle to be well tolerated, with no product-related serious adverse events in >200 treated subjects.

Objectives:

Primary

-To determine the safety and tolerability of escalating doses of a heat-killed yeast-based vaccine that targets tumors that express CEA.

Secondary

* To evaluate CD4 and CD8 immunologic response as measured by an increase in CEA-specific T cells measured by ELISPOT in HLA-A2, -A3 and -A24(+) patients, and proliferation in response to CEA protein.
* To evaluate evidence of clinical benefit, such as progression-free survival, RECIST criteria, reduction in serum markers, and/or reduction in circulating tumor cells.

Eligibility: (dose escalation phase)

Must have metastatic cancer that is CEA-positive (either a CEA serum level > 5 ng/mL or a tumor that stains positive for CEA in > 20% of a tumor block).

Must have completed or had disease progression on at least one prior line of disease-appropriate therapy, or not be a candidate for therapy of proven efficacy for their disease.

Must be ECOG Performance Status 0 2.

Should have no autoimmune diseases; no evidence of immune dysfunction; no serious intercurrent medical illness;

No untreated brain metastasis (or local treatment of brain metastases within the last 6 months)

Any hypersensitivity reaction to yeast-based products.

Eligibility: (extension phase: 10 additional patients at highest tested dose/MTD)

Same as for the dose escalation phase with the following exceptions:

* Patients must be HLA-A2, -A3, or -A24(+) for immunologic monitoring
* ECOG PS = 0 1

Design:

This is an open label, phase I trial with sequential cohorts of patients (3-6 patients per dose cohort) with dose escalation of heat-killed GI-6207 vaccine (see statistical analysis section).

GI 6207 vaccine will be administered subcutaneously at 4 sites biweekly for 7 visits (days 1, 15, 29, 43, 57, 71, 85), then monthly until patients meet off-study criteria.

All patients on a given dose level will have completed 1 month on-study before enrollment can begin on the next dose level or on the extension phase (see statistical analysis section).

ELIGIBILITY:
* INCLUSION CRITERIA:

A. Histologically confirmed carcinoma by the NIH Laboratory of Pathology that has been shown to express CEA (either a CEA serum level > 5 microg/L or a tumor that stains positive for CEA in > 20% of a tumor block).

B. Completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease, or not be a candidate for therapy of proven efficacy for their disease.

C. 18 years of age or greater.

D. Must have metastatic disease that is measurable or non-measurable but evaluable (e.g., pleural effusion or present on bone scan).

E. Ability to understand and the willingness to sign a written informed consent document.

F. ECOG performance status of 0 2 (Karnofsky greater than or equal to 50).

G. Serum creatinine less than or equal to 1.5 times upper limit of normal OR creatinine clearance on a 24-h urine collection of greater than or equal to 60 mL/min.

H. ALT and AST less than or equal to 2.5 times the upper limits of normal.

I. Total bilirubin less than or equal to 1.5 times upper limit of normal OR in patients with Gilbert s syndrome, a total bilirubin less than or equal to 3.0.

J. Recovered completely from any reversible toxicity associated with recent therapy. Typically this is 3 4 weeks for patients who most recently received cytotoxic therapy, except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery. There should be a minimum of 2 weeks from any prior chemotherapy, immunotherapy and/or radiation.

K. Hematological eligibility parameters (within 16 days of starting therapy):

* Granulocyte count greater than or equal to 1,500/mm(3)
* Platelet count greater than or equal to 100,000/mm(3)

L. Prior immune therapy (e.g. related vaccinia and fowlpox vaccines or antigen-specific peptides) is allowed.

M. Men and women must agree to use effective birth control or abstinence during and for a period of 4 months after the last vaccination therapy.

N. Patients with prostate cancer must continue to receive GnRH agonist therapy (unless orchiectomy has been done).

O. Patients must be negative for yeast allergy skin test.

P. Patients must have baseline pulse oximetry greater than 90% on room air.

INCLUSION CRITERIA (EXTENSION PHASE: 10 ADDITIONAL PATIENTS AT HIGHEST TESTED DOSE/MTD):

Eligibility: Same as with the dose escalation phase with the following exceptions:

* Patients must be HLA-A2, A3, or A24 positive for immunologic monitoring.
* ECOG PS equal to 0 1.

EXCLUSION CRITERIA:

A. Patients should have no evidence of immune dysfunction as listed below.

* Human immunodeficiency virus positivity due to the potential for decreased immune response to the vaccine.
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. Patients with endocrine autoimmune disease that is controlled by replacement therapy, including thyroid disease and adrenal disease; or those with vitiligo, may be enrolled.
* Concurrent use of systemic steroids, except for physiologic doses for systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids to prevent IV contrast, allergic reaction, or anaphylaxis (in patients who have known contrast allergies) are allowed.

B. History of allergy or untoward reaction to yeast-based products (any hypersensitivity to yeast-based products will be excluded).

C. Pregnant or breast-feeding women.

E. Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.

F. Untreated brain metastases (or local treatment of brain metastases within the last 6 months) due to the poor prognosis of these patients and difficulty ascertaining the cause of neurologic toxicities.

G. Concurrent chemotherapy. An exception is to allow for patients on the extension phase only with breast cancer who are receiving trastuzumab to continue therapy with trastuzumab while receiving the vaccine treatment.

K. Chronic hepatitis infection, including B and C, because of potential immune impairment.

L. Patients requiring continuous tricyclic antidepressant therapy should be excluded due to the interference with the yeast skin test in creating false negative test results.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-03-13; Study Completion 2012-08-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of escalating doses of a heated-killed yeast-based vaccine that targets tumors that express CEA.

SECONDARY OUTCOMES:
To evaluate CD4 and CD8 immunologic response. To evaluate humoral immune response to yeast antigen. To evaluate evidence of clinical benefit such as PFS, OR, & decreases in circulating tumor cells & tumor markers.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Robbins PF, Eggensperger D, Qi CF, Schlom J. Definition of the expression of the human carcinoembryonic antigen and non-specific cross-reacting antigen in human breast and lung carcinomas. Int J Cancer. 1993 Apr 1;53(6):892-7. doi: 10.1002/ijc.2910530604. PMID 8386136
- [Background] Kass ES, Greiner JW, Kantor JA, Tsang KY, Guadagni F, Chen Z, Clark B, De Pascalis R, Schlom J, Van Waes C. Carcinoembryonic antigen as a target for specific antitumor immunotherapy of head and neck cancer. Cancer Res. 2002 Sep 1;62(17):5049-57. PMID 12208760
- [Background] Hodge JW, Tsang KY, Poole DJ, Schlom J. General keynote: vaccine strategies for the therapy of ovarian cancer. Gynecol Oncol. 2003 Jan;88(1 Pt 2):S97-104; discussion S110-3. doi: 10.1006/gyno.2002.6694. No abstract available. PMID 12586096